CLINICAL TRIAL: NCT00511316
Title: A Randomized Placebo-Controlled Trial of Montelukast in Maintenance Therapy of Asymptomatic Eosinophilic Esophagitis
Brief Title: Trial of Montelukast in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-003373
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Experimental): 20 mg montelukast daily for 6 months
  Interventions: Drug: Montelukast/ Singulair
- Placebo (Placebo Comparator): 20 mg daily placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast/ Singulair — 20 mg daily for six months
  Other Names: Singulair
  Arms: Drug
Drug: Placebo — Placebo 20 mg daily for 6 months
  Arms: Placebo

SUMMARY:
Evaluate clinical effectiveness of oral montelukast compared to placebo on prevention of dysphagia and food impaction in patients with EE.

Also evaluate tolerance and safety of oral montelukast in treatment of EE.

DETAILED DESCRIPTION:
We will randomize in a double blind manner 60 consecutive consenting patients being evaluated at the three Mayo Clinic Medical Centers with EE to montelukast 20mg daily or placebo daily for six months? time. Patients will be in remission after treatment with topical fluticasone therapy before enrollment. Patients will fill out a validated dysphagia and side effect questionnaire before, during, and at the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* > 14 eosinophils / hpf on biopsies from mid esophagus within the 6 months.
* Abnormal dysphagia questionnaire (Question 1a yes, question 1c >/= mild and question 2 >/= less than once a week) prior to topical steroid treatment. This questionnaire has recently been validated.
* Normal dysphagia questionnaire after topical steroid treatment (Having an answer of no to question 1a: Have you had trouble swallowing, not associated with other cold symptoms? over the past two weeks since having completed the swallowed steroid treatment).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
evaluate effectiveness of oral montelukast in treatment of EE. | 6 months

SECONDARY OUTCOMES:
evaluate safety of montelukast in eosinophilic esophagitis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Alexander, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Alexander JA, Ravi K, Enders FT, Geno DM, Kryzer LA, Mara KC, Smyrk TC, Katzka DA. Montelukast Does not Maintain Symptom Remission After Topical Steroid Therapy for Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2017 Feb;15(2):214-221.e2. doi: 10.1016/j.cgh.2016.09.013. Epub 2016 Sep 17. PMID 27650328